CLINICAL TRIAL: NCT07267000
Title: Exercise as a Tool to Improve Response to Immunotherapy in Non-small Cell Lung Cancer
Acronym: ImmuEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: University of Graz (Other); Austrian Science Fund (FWF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ImmuEX; PAT1625724 (Other: FWF Austrian Sience Fund)
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer; Exercise Training; Immunotherapy
Keywords: Non-small cell lung cancer; Exercise; Immunotherapy; Outcome
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous Exercise (Experimental): Patients in this arm will undergo a 12-week training therapy regimen consisting of twice weekly supervised moderate-intensity continuous exercise (MICE) and home-based walking exercise for 30 minutes, five times a week, in addition.
  Interventions: Behavioral: Exercise
- High Intensity Interval Exercise (Experimental): Patients in this arm will undergo a 12-week training therapy regimen consisting of twice weekly supervised high-intensity interval exercise and home-based walking exercise for 30 minutes, five times a week, in addition.
  Interventions: Behavioral: Exercise
- Controls (Active Comparator): Patients in this arm will receive general recommendations on an active lifestyle, but will not take part in supervised training sessions and are not asked to do home-based exercise either.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Exercise — 1 study arm doing continuous type exercise will be compared to 1 study arm doing high-intensity interval exercise, over the course of 12 weeks, respectively. Both arms will be compared to sedentary control patients.
  Other Names: Home-based walking exercise
  Arms: Continuous Exercise; High Intensity Interval Exercise
Other: Control — For patients in the control group, general exercise recommendations (e.g. recommendations by the CDC suitable for all adult individuals) will be given, however, no training therapy intervention is done and no home-based walking exercise is required either.
  Arms: Controls

SUMMARY:
This project is about the effect of a 12-week training therapy intervention in patients suffering from non-small cell lung cancer. It has widely been accepted that exercise is preventive against certain types of cancer. Individuals following an active lifestyle have a significantly lower risk for several chronic diseases, including cancer, as compared to sedentary ones. However, evidence is still lacking for exercise as part of routine cancer treatment (as it has already been implemented routinely in patients with heart disease, for example). In this study, patients suffering from non-small cell lung cancer undergo either a 12-week training program consisting of moderate-intensity continuous exercise (MICE), or a 12-week program with high-intensity interval exercise. Both groups will be compared to a control group receiving standard exercise recommendations. The response to immunotherapy, measured by the radiologic therapy response, will be the main endpoint. Additionally, blood will be taken from the patients at different timepoints, and blood samples will be tested for immunologic changes. FACS analysis will be used to assess the properties of immune cells and potential changes upon the exercise regimen. Mitochondrial function will be assessed via the Seahorse machine, and mass spectrometry (lipidomics) will be used for the analysis of lipid profile changes.

DETAILED DESCRIPTION:
Lung cancer is the number one cause of cancer-related deaths worldwide. A few decades ago, the prognosis at lung cancer first diagnosis was generally poor with only a few months of median survival. New immunotherapy treatment regimens have markedly improved survival times - especially in certain histologic and molecular pathologic subtypes. The positive effect of exercise on the incidence of several cancer entities such as colorectal- or breast cancer, has been demonstrated previously. Physically active individuals are diagnosed with cancer significantly less often as compared to sedentary people. In oncologic follow-up care, a positive effect of exercise and training with an advantage in survival has also been proven, e.g. in breast cancer patients.

In addition, existing data shows a positive effect of exercise on the immune system: active individuals show a different pattern of proinflammatory markers in the blood serum, with every exercise session generating an immune-stimulatory effect which changes the immunologic serum profile also at rest. Thus, regular exercise has an anti-inflammatory long-term effect.

Hypothesis and Objectives: With our project we seek to demonstrate a possible benefit on immunotherapy response upon a medically guided training regimen.

Setting and Methods. To exactly define "exercise" in this setting, as a first step we will test two exercise types in healthy individuals. According to their individual exercise capacity as determined by spiroergometry, healthy subjects will either perform moderate-intensity continuous exercise (MICE), or a high-intensity interval training (HIIT). By means of venous blood sampling before and after training we shall determine the respective changes of serum immune markers through exercise. The same two training types will then be performed by lung cancer patients upon immunotherapy, with one patient group doing MICE-sessions, one group doing the HIIT and a third group who will receive general exercise recommendations. Response to therapy and inflammatory serum parameters will be compared between the groups. Exercising patients will be advised to train once a week under medical supervision, and to walk briskly for 30 minutes every day of the week in addition. Our hypothesis is, that exercise should be implemented as a complementary treatment strategy in every oncologic therapy setting, possibly improving not only physical health and wellbeing but also treatment response. In addition to improving the patients' quality of life by a better physical capacity and fitness, helping them in their everyday activities, we propose that the implementation of exercise programs in various oncologic settings in future may improve the patients' outcome.

Scientific Novelty. Standardization of exercise regimens in oncologic scenarios in the existing literature is generally poor. We carry out one of the few studies where the type, duration, timing and intensity of exercise in both exercise groups is clearly defined, comparing two different training types to sedentary control patients, respectively. Exercise needs to be seen as a drug, and like in any drug the optimum dose must be clearly outlined. Moreover, we will implement a priming exercise in our study, meaning that patients exercise close to the administration of immunotherapy, hypothesizing that this may further ameliorate therapy response.

ELIGIBILITY:
Inclusion Criteria: Patients suffering from non-small cell lung cancer of any histologic subtype at first diagnosis, receiving a treatment regimen comprising immunotherapy (with or without chemotherapy).

-

Exclusion Criteria:

* Kachexia (BMI<18.5)
* instable bone metastases
* orthopedic condition rendering the patient unable to ride a stationary bike
* any medical contraindication for exercise and training

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Response to immunotherapy | From enrollment to the first CT scan after the 12 week training therapy intervention
  Response to immunotherapy will be measured on the one hand metrically based on the change of tumor volume in mm3, and on the other hand based on the RECIST criteria.

SECONDARY OUTCOMES:
Immunologic changes - FACS analysis | From enrollment to after completion of the 12 week training therapy intervention
  The proportion of immune cell subtypes will be determined by means of FACS analysis before and after the exercise intervention.
Seahorse analysis | From enrollment to after completion of the exercise intervention
  "Seahorse analysis" refers to a biological assay, conducted using a Seahorse XF Analyzer from Agilent, that measures the real-time metabolic activity of live cells by simultaneously assessing mitochondrial respiration and glycolysis. The assay does this by measuring two key parameters: the oxygen consumption rate (OCR), which indicates mitochondrial respiration, and the extracellular acidification rate (ECAR), which is linked to glycolysis. It is used to understand changes in cellular energy production, stress responses, oxygen consumption and proton production.
Mass spectrometry - Lipidomics | From enrollment to after completion of the 12 week exercise intervention.
  Lipidomics is used to describe the complete lipid profile within the patients' immune cells. It is a subset of the "metabolome". As opposed to classic analysis of carbohydrate metabolism, lipids are more stable, allowing for an analysis of frozen PBMCs. Our hypothesis is that upon the exercise program, lipidomics of the immune cells significantly change, allowing for a more favorable antitumor immune response.
Cytokine profiling | From enrollment to after completion of the 12 week training therapy intervention.
  The distribution (increases) in proinflammatory cytokines will be measured before and after the 12 week exercise intervention. In addition, the cytokine serum profile changes immediately after an exercise bout will be measured as well, based on blood sampling. Cytokines will be analysed with an ELISA kit, focusing on cytokine subsets usually affected by exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided
It depends on the data that is measured, especially as far as the basic research experiments (FACS, Seahorse, Cytokines, Lipidomics) are concerned. If the data is promising, we might share it with other researchers for additional publication.

REFERENCES:
- [Background] Martin-Ruiz A, Fiuza-Luces C, Rincon-Castanedo C, Fernandez-Moreno D, Galvez BG, Martinez-Martinez E, Martin-Acosta P, Coronado MJ, Franco-Luzon L, Gonzalez-Murillo A, Ramirez M, Provencio M, Lucia A. Benefits of exercise and immunotherapy in a murine model of human non-small-cell lung carcinoma. Exerc Immunol Rev. 2020;26:100-115. PMID 32139351
- [Background] Ungvari Z, Fekete M, Varga P, Munkacsy G, Fekete JT, Lehoczki A, Buda A, Kiss C, Ungvari A, Gyorffy B. Exercise and survival benefit in cancer patients: evidence from a comprehensive meta-analysis. Geroscience. 2025 Jun;47(3):5235-5255. doi: 10.1007/s11357-025-01647-0. Epub 2025 Apr 12. PMID 40220151
- [Background] Winters-Stone KM, Neil SE, Campbell KL. Attention to principles of exercise training: a review of exercise studies for survivors of cancers other than breast. Br J Sports Med. 2014 Jun;48(12):987-95. doi: 10.1136/bjsports-2012-091732. Epub 2013 Jan 4. PMID 23293010
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Rezende LFM, Sa TH, Markozannes G, Rey-Lopez JP, Lee IM, Tsilidis KK, Ioannidis JPA, Eluf-Neto J. Physical activity and cancer: an umbrella review of the literature including 22 major anatomical sites and 770 000 cancer cases. Br J Sports Med. 2018 Jul;52(13):826-833. doi: 10.1136/bjsports-2017-098391. Epub 2017 Nov 16. PMID 29146752
- [Background] Ashcraft KA, Peace RM, Betof AS, Dewhirst MW, Jones LW. Efficacy and Mechanisms of Aerobic Exercise on Cancer Initiation, Progression, and Metastasis: A Critical Systematic Review of In Vivo Preclinical Data. Cancer Res. 2016 Jul 15;76(14):4032-50. doi: 10.1158/0008-5472.CAN-16-0887. Epub 2016 Jul 5. PMID 27381680
- Available data/document: Individual Participant Data Set — https://project-redcap.org/ — IPD will be collected in the REDCap database. Since enrolment of patients has not started yet, no data has yet been entered. We are undecided on whether to share IPD with other researchers in future.